CLINICAL TRIAL: NCT06554925
Title: SEx-specific Differences in Cardiac Surgery Patients (SECS). A Retrospective Registration and Evaluation of Characteristics and Perioperative Management of Cardiac Surgery Patients
Brief Title: SEx-specific Differences in Cardiac Surgery Patients (SECS).
Acronym: SECS
Status: Recruiting | Type: Observational
Sponsor: Jennifer Breel (Other)
Responsible Party: Sponsor-Investigator, Jennifer Breel, Research coordinator, Amsterdam University Medical Centers (UMC), Location Academic Medical Center (AMC)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Other Study IDs: W22_050 # 22.081
Record Dates: First submitted 2022-03-20; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Female; Male; Surgery, Cardiac
Keywords: anesthesia; sex-specific differences; cardiac surgery; care pathways
MeSH Terms: interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Female: Female sex undergoing cardiac surgery
  Interventions: Procedure: Cardiac surgery
- Male: Male sex undergoing cardiac surgery
  Interventions: Procedure: Cardiac surgery

INTERVENTIONS:
Procedure: Cardiac surgery — The difference in males and females undergoing cardiac surgery of all types

SUMMARY:
The aim of this study is to evaluate the differences between females and males undergoing cardiac surgery. The investigators will look at perioperative factors such as adaption of body weight, previous medical history, pharmacokinetics, transfusion, coagulation, cardiopulmonary bypass (CPB) related factors, cardiac function, inotropic requirements, risk, and outcome scores as well as morbidity and mortality at sort-term (within 30 days) and long-term (90 days and 1 year).

DETAILED DESCRIPTION:
There are now an increasing number of studies on preoperative cardiovascular differences in females and males, but no study to date has focused on a female-specific approach to perioperative anaesthesia and critical care in cardiac surgery patients.

Given the higher mortality and morbidity in females after cardiac surgery, as well as the abovementioned sex differences, it is likely that females require different perioperative care than males, for better and faster recovery.

The investigators hypothesise that females require different perioperative care (pathways) compared to males when undergoing cardiac surgery. The investigators would therefore like to investigate which factors are different in female and male patients, by setting up a database of perioperative parameters. By identifying the factors that adversely affect morbidity and mortality in females and linking these parameters, the investigators would like to improve outcome in fmales after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years
* All patients who underwent cardiac surgery from 1 January 1998 in the AUMC, location VUmc, until 1 June 2021.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of male and female patients, 18 years and older. The study group consists of all patients who underwent cardiothoracic surgery from 1998 in the AUMC, location VUmc until June 2021. Observational retrospective data collection from the mandatory Quality Assurance database of the Netherlands Heart Registry, supplemented with data from the electronic patient files (EPIC).
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2030-03-01 (Estimated); Study Completion 2031-03-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative mortality | Measured at 20 years postoperatively
  Incidence of perioperative mortality
Postoperative mortality | Measured at 30 days postoperatively
  Incidence of perioperative mortality
Postoperative mortality | Measured at 1 year postoperatively
  Incidence of perioperative mortality
Postoperative mortality | Measured at 5 years postoperatively
  Incidence of perioperative mortality

SECONDARY OUTCOMES:
Postoperative complications (Morbidity) | Measured at 30 days
  Incidence of peroperative and post-operative complications
Postoperative complications (Morbidity) | Measured at 90 days
  Incidence of peroperative and post-operative complications
Postoperative complications (Morbidity) | Measured at 365 days
  Incidence of peroperative and post-operative complications
Development of a predictive risk score using a composite outcome | Up to 30 days postoperatively
  Predictive risk score

CONTACTS AND LOCATIONS:
Overall Officials: Markus W Hollmann, Professor, Principal Investigator — Anesthesiology and Pain Medicine, Amsterdam Medical Center
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cho L, Kibbe MR, Bakaeen F, Aggarwal NR, Davis MB, Karmalou T, Lawton JS, Ouzounian M, Preventza O, Russo AM, Shroyer AW, Zwischenberger BA, Lindley KJ. Cardiac Surgery in Women in the Current Era: What Are the Gaps in Care? Circulation. 2021 Oct 5;144(14):1172-1185. doi: 10.1161/CIRCULATIONAHA.121.056025. Epub 2021 Oct 4. PMID 34606298
- [Background] Dixon LK, Di Tommaso E, Dimagli A, Sinha S, Sandhu M, Benedetto U, Angelini GD. Impact of sex on outcomes after cardiac surgery: A systematic review and meta-analysis. Int J Cardiol. 2021 Nov 15;343:27-34. doi: 10.1016/j.ijcard.2021.09.011. Epub 2021 Sep 11. PMID 34520795
- [Background] Nanegrungsunk D, Patel S, Jan T, Ngai JY. Preoperative Care Practice for Female Cardiac Patients: A Survey From the Society of Cardiovascular Anesthesiologists. J Cardiothorac Vasc Anesth. 2022 Mar;36(3):920-921. doi: 10.1053/j.jvca.2021.09.054. Epub 2021 Oct 3. No abstract available. PMID 34776353
- [Background] Peters SAE, Kluin J. Why do women do worse after coronary artery bypass grafting? Eur Heart J. 2021 Dec 28;43(1):29-31. doi: 10.1093/eurheartj/ehab617. No abstract available. PMID 34524421